CLINICAL TRIAL: NCT06115720
Title: CIA: Consent in Anaesthesia, Prospective Randomised-controlled Trial
Brief Title: Consent in Anaesthesia
Acronym: CIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 305199; 23SM8319 (Other: Imperial College Healthcare NHS Trust)
Record Dates: First submitted 2023-10-19; First posted 2023-11-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Regional Anesthesia; Patient Satisfaction
Keywords: Consent; Patient information; Regional Anaesthesia; General Anaesthesia
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Recruited participants, randomised to one of two groups. Control group: standard video verbal consent process for GA and RA for orthopaedic surgery. This verbal communication will be pre-recorded and shown to the participant.
  Intervention group: Same pre-recorded standard verbal consent, additionally recorded video of the anaesthetic process for both GA and RA.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcome assessors are blinded to which arm the participants are allocated when analysing the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard video verbal consent process (No Intervention): The control group will undergo the standard video verbal consent process for both GA and RA for orthopaedic surgery. This will be delivered using a standardised video script that will be generated from existing certified material.
- Video assisted consent process (Experimental): The intervention group will also be shown the same pre-recorded standard verbal consent, but following this will additionally be shown a specifically recorded video of the anaesthetic process for both GA and RA.
  Interventions: Other: Video assisted consent

INTERVENTIONS:
Other: Video assisted consent — The intervention group will also be shown the same pre-recorded standard verbal consent, but following this will additionally be shown a specifically recorded video of the anaesthetic process for both GA and RA. This video will aim to communicate the same information as that found in the traditional verbal consent, using an actor undergoing an anaesthetic to provide context.
  Arms: Video assisted consent process

SUMMARY:
DESIGN: Prospective randomised-controlled trial AIM: To determine whether presenting both techniques of general anaesthesia and regional anaesthesia in an unbiased manner, with video media, aids the anaesthetic consent process, compared to standard verbal consent alone.

OUTCOME MEASURES

Primary outcome:

- Participants' satisfaction regarding the anaesthetic consent process

Secondary outcomes:

* Knowledge, attitudes and practices towards anaesthesia
* Participants' choice of anaesthetic technique POPULATION: General adult population (>18yrs), males and females DURATION: 2 years

DETAILED DESCRIPTION:
The main aim of this study is to determine if presenting both anaesthetic techniques of general anaesthesia (GA) and regional anaesthesia (RA) to a participant in an unbiased manner, with video media, affects the participants' satisfaction, knowledge of, and attitudes towards anaesthesia. The investigators hypothesise that using video media will improve participants' satisfaction with the anaesthetic consent process, thereby resulting in better quality informed consent.

Participant's knowledge retention, attitudes and practices towards GA and RA, measured by an knowledge, attitudes and practices (KAP) questionnaire based on the consent process. Participant's stated preference for anaesthetic technique (i.e. General or Regional).

Several studies have shown that video-based patient education have led to better patient comprehension and satisfaction as well as reduced patient anxiety during the consent process compared to verbal consent.

Examples The use of portable video media vs standard verbal communication in the urological consent process: a multicentre, randomised controlled, crossover trial showed that 80.7% of patients preferred portable video media (PVM) and 19.3% preferred standard video consent (SVC). PVM improves patient's understanding compared with SVC and is a more effective means of content delivery to patients in terms of overall preference and knowledge gained during the consent process.

Effect of preoperative multimedia information on perioperative anxiety in patients undergoing procedures under regional anaesthesia, showed that preoperative multimedia information reduces the anxiety of patients undergoing surgery under regional anaesthesia. This type of information is easily delivered and can benefit many patients.

Oxford Video Informed Consent Tool (OxVIC): a pilot study of informed video consent in spinal surgery and preoperative patient satisfaction concluded: "Introduction of a video consent tool was found to be a positive adjunct to traditional consenting methods. Patient-clinician consent dialogue can now be documented. A randomised controlled study to further evaluate the effects of video consent on patients' retention of information, preoperative and postoperative anxiety, patient reported outcome measures as well as length of stay may be beneficial."

During the Covid pandemic, with the need for social distancing, this is particularly useful and allows for involvement of family support for decision making by allowing sufficient time for informed consent to be made.

The aim of this study is to determine if the use of video assisted consent during the anaesthetic consent process, for both GA and RA, affects the participants' satisfaction, knowledge of, and attitudes towards, anaesthesia.

The investigators hypothesise that using video media will improve participant knowledge, understanding and satisfaction of the anaesthetic consent process, thereby resulting in better quality informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to pre-operative orthopaedic surgical clinic
* Informed consent

Exclusion Criteria:

* Patients <18 years or vulnerable groups
* Inability to communicate in English or language difficulty that requires an interpreter
* Severe vision or hearing loss if lack of other communication channels
* Private patients
* Prisoners
* Patients who reside outside the United Kingdom (home address)
* Opt-out patients on General Practitioner register

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction CSQ-8 | 5 -10 minutes
  Client Satisfaction Questionnaire is a questionnaire measuring satisfaction. Response options differ from item to item, but all are based on a four-point scale. Examples include: "How satisfied are you with the amount of help you have received?" (which response options: 1 = "Quite dissatisfied", 2 = "Indifferent or mildly dissatisfied", 3 = "Mostly satisfied", 4 = "Very satisfied"; and, "Have the services you received helped you to deal more effectively with your problems?" (Which has the response options: 4 = Yes, they helped a great deal", 3 = "Yes, they helped somewhat", 2 = "No, they didn't help", 1 = "No, they seemed to make things worse". with an overall score is produced by summing all item responses. For the CSQ-8 version, scores range from 8 to 32, with higher values indicating higher satisfaction.

SECONDARY OUTCOMES:
KAP Questionnaire | 5 - 10 minutes
  Knowledge, attitudes and practices towards anaesthesia. Response options differ from item to item, but all are based on a five-point scale. Examples include: "How afraid are you of a sore throat?" (which response options: 1 = "Very unafraid", 2 = "Unafraid", 3 = "Neither afraid or unafraid", 4 = "Afraid", 5 = "Very Afraid"; and, "Having permanent nerve damage" (Which has the response options: 1 = "Very unafraid", 2 = "Unafraid", 3 = "Neither afraid or unafraid", 4 = "Afraid", 5 = "Very Afraid"; with an overall score is produced by summing all item responses. Higher values indicating a higher level of being afaid.
Anaesthetic choice | 1 - 2 minutes
  Participants' preferred choice choice of anaesthetic technique: General or Regional tick box

CONTACTS AND LOCATIONS:
Overall Officials: Boyne Bellew, Principal Investigator — Imperial College Healthcare NHS Trust; Christopher Mullington, Principal Investigator — Imperial College Healthcare NHS Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woodall NM, Cook TM. National census of airway management techniques used for anaesthesia in the UK: first phase of the Fourth National Audit Project at the Royal College of Anaesthetists. Br J Anaesth. 2011 Feb;106(2):266-71. doi: 10.1093/bja/aeq339. Epub 2010 Dec 4. PMID 21131655
- [Background] Sury MR, Palmer JH, Cook TM, Pandit JJ. The state of UK anaesthesia: a survey of National Health Service activity in 2013. Br J Anaesth. 2014 Oct;113(4):575-84. doi: 10.1093/bja/aeu292. Epub 2014 Aug 7. PMID 25236896
- [Background] O'Donnell BD, Ryan H, O'Sullivan O, Iohom G. Ultrasound-guided axillary brachial plexus block with 20 milliliters local anesthetic mixture versus general anesthesia for upper limb trauma surgery: an observer-blinded, prospective, randomized, controlled trial. Anesth Analg. 2009 Jul;109(1):279-83. doi: 10.1213/ane.0b013e3181a3e721. PMID 19535722
- [Background] Galos DK, Taormina DP, Crespo A, Ding DY, Sapienza A, Jain S, Tejwani NC. Does Brachial Plexus Blockade Result in Improved Pain Scores After Distal Radius Fracture Fixation? A Randomized Trial. Clin Orthop Relat Res. 2016 May;474(5):1247-54. doi: 10.1007/s11999-016-4735-1. Epub 2016 Feb 11. PMID 26869374
- [Background] Mulroy MF, Larkin KL, Batra MS, Hodgson PS, Owens BD. Femoral nerve block with 0.25% or 0.5% bupivacaine improves postoperative analgesia following outpatient arthroscopic anterior cruciate ligament repair. Reg Anesth Pain Med. 2001 Jan-Feb;26(1):24-9. doi: 10.1053/rapm.2001.20773. PMID 11172507
- [Background] Williams BA, Bottegal MT, Kentor ML, Irrgang JJ, Williams JP. Rebound pain scores as a function of femoral nerve block duration after anterior cruciate ligament reconstruction: retrospective analysis of a prospective, randomized clinical trial. Reg Anesth Pain Med. 2007 May-Jun;32(3):186-92. doi: 10.1016/j.rapm.2006.10.011. PMID 17543812
- [Background] Bulka CM, Shotwell MS, Gupta RK, Sandberg WS, Ehrenfeld JM. Regional anesthesia, time to hospital discharge, and in-hospital mortality: a propensity score matched analysis. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):381-6. doi: 10.1097/AAP.0000000000000121. PMID 25025697
- [Background] Yentis SM, Hartle AJ, Barker IR, Barker P, Bogod DG, Clutton-Brock TH, Ruck Keene A, Leifer S, Naughton A, Plunkett E. AAGBI: Consent for anaesthesia 2017: Association of Anaesthetists of Great Britain and Ireland. Anaesthesia. 2017 Jan;72(1):93-105. doi: 10.1111/anae.13762. PMID 27988961
- [Background] Winter M, Kam J, Nalavenkata S, Hardy E, Handmer M, Ainsworth H, Lee WG, Louie-Johnsun M. The use of portable video media vs standard verbal communication in the urological consent process: a multicentre, randomised controlled, crossover trial. BJU Int. 2016 Nov;118(5):823-828. doi: 10.1111/bju.13595. Epub 2016 Aug 25. PMID 27440499
- [Background] Armstrong AW, Alikhan A, Cheng LS, Schupp C, Kurlinkus C, Eisen DB. Portable video media for presenting informed consent and wound care instructions for skin biopsies: a randomized controlled trial. Br J Dermatol. 2010 Nov;163(5):1014-9. doi: 10.1111/j.1365-2133.2010.10067.x. PMID 20977443
- [Background] Jlala HA, French JL, Foxall GL, Hardman JG, Bedforth NM. Effect of preoperative multimedia information on perioperative anxiety in patients undergoing procedures under regional anaesthesia. Br J Anaesth. 2010 Mar;104(3):369-74. doi: 10.1093/bja/aeq002. Epub 2010 Feb 1. PMID 20124283
- [Background] Mawhinney G, Thakar C, Williamson V, Rothenfluh DA, Reynolds J. Oxford Video Informed Consent Tool (OxVIC): a pilot study of informed video consent in spinal surgery and preoperative patient satisfaction. BMJ Open. 2019 Jul 24;9(7):e027712. doi: 10.1136/bmjopen-2018-027712. PMID 31345967
- [Background] Zhang Y, Ruan X, Tang H, Yang W, Xian Z, Lu M. Video-Assisted Informed Consent for Cataract Surgery: A Randomized Controlled Trial. J Ophthalmol. 2017;2017:9593631. doi: 10.1155/2017/9593631. Epub 2017 Jan 16. PMID 28191349
- [Background] Tipotsch-Maca SM, Varsits RM, Ginzel C, Vecsei-Marlovits PV. Effect of a multimedia-assisted informed consent procedure on the information gain, satisfaction, and anxiety of cataract surgery patients. J Cataract Refract Surg. 2016 Jan;42(1):110-6. doi: 10.1016/j.jcrs.2015.08.019. PMID 26948785
- [Background] Batuyong ED, Jowett AJ, Wickramasinghe N, Beischer AD. Using multimedia to enhance the consent process for bunion correction surgery. ANZ J Surg. 2014 Apr;84(4):249-54. doi: 10.1111/ans.12534. PMID 24812709
- [Background] Rossi MJ, Guttmann D, MacLennan MJ, Lubowitz JH. Video informed consent improves knee arthroscopy patient comprehension. Arthroscopy. 2005 Jun;21(6):739-43. doi: 10.1016/j.arthro.2005.02.015. PMID 15944633
- [Background] Eggers C, Obliers R, Koerfer A, Thomas W, Koehle K, Hoelscher AH, Bollschweiler E. A multimedia tool for the informed consent of patients prior to gastric banding. Obesity (Silver Spring). 2007 Nov;15(11):2866-73. doi: 10.1038/oby.2007.340. PMID 18070779
- [Background] Bowers N, Eisenberg E, Montbriand J, Jaskolka J, Roche-Nagle G. Using a multimedia presentation to improve patient understanding and satisfaction with informed consent for minimally invasive vascular procedures. Surgeon. 2017 Feb;15(1):7-11. doi: 10.1016/j.surge.2015.09.001. Epub 2015 Oct 14. PMID 26464072
- [Background] Celik EC, Ekinci M, Ciftci B, Golboyu BE, Kilinc OO. Influence of visual information on consent for invasive procedures in intensive care unit. Niger J Clin Pract. 2018 May;21(5):609-613. doi: 10.4103/njcp.njcp_437_16. PMID 29735862
- [Background] Groves ND, Humphreys HW, Williams AJ, Jones A. Effect of informational internet web pages on patients' decision-making: randomised controlled trial regarding choice of spinal or general anaesthesia for orthopaedic surgery. Anaesthesia. 2010 Mar;65(3):277-82. doi: 10.1111/j.1365-2044.2009.06211.x. PMID 20336817
- [Background] Elkassabany NM, Abraham D, Huang S, Kase B, Pio F, Hume E, Israelite C, Liu J. Patient education and anesthesia choice for total knee arthroplasty. Patient Educ Couns. 2017 Sep;100(9):1709-1713. doi: 10.1016/j.pec.2017.04.014. Epub 2017 Apr 29. PMID 28487116
- [Background] Zarnegar R, Brown MR, Henley M, Tidman V, Pathmanathan A. Patient perceptions and recall of consent for regional anaesthesia compared with consent for surgery. J R Soc Med. 2015 Nov;108(11):451-6. doi: 10.1177/0141076815604494. Epub 2015 Oct 2. PMID 26432814
- [Background] Salzwedel C, Petersen C, Blanc I, Koch U, Goetz AE, Schuster M. The effect of detailed, video-assisted anesthesia risk education on patient anxiety and the duration of the preanesthetic interview: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):202-9, table of contents. doi: 10.1213/01.ane.0000287665.96156.72. PMID 18165579
- [Background] Mihalj M, Carrel T, Gregoric ID, Andereggen L, Zinn PO, Doll D, Stueber F, Gabriel RA, Urman RD, Luedi MM. Telemedicine for preoperative assessment during a COVID-19 pandemic: Recommendations for clinical care. Best Pract Res Clin Anaesthesiol. 2020 Jun;34(2):345-351. doi: 10.1016/j.bpa.2020.05.001. Epub 2020 May 14. PMID 32711839
- [Background] Kickbusch IS. Health literacy: addressing the health and education divide. Health Promot Int. 2001 Sep;16(3):289-97. doi: 10.1093/heapro/16.3.289. PMID 11509466
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Rowlands G, Khazaezadeh N, Oteng-Ntim E, Seed P, Barr S, Weiss BD. Development and validation of a measure of health literacy in the UK: the newest vital sign. BMC Public Health. 2013 Feb 7;13:116. doi: 10.1186/1471-2458-13-116. PMID 23391329

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT06115720/Prot_SAP_000.pdf